CLINICAL TRIAL: NCT06836440
Title: The Impact of Spectacle Intervention for Refractive Error and Presbyopia on Cognitive Function in Rural Older Adults
Brief Title: Impact of Glasses for Vision Problems on Cognitive Function in Rural Older Adults
Acronym: CLEVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuju Wu (Other)
Responsible Party: Sponsor-Investigator, Yuju Wu, Associate Professor, Sichuan University
Organization: Sichuan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Gwll202464
Record Dates: First submitted 2025-02-12; First posted 2025-02-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cognition Disorders
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Prescription Glasses Intervention group (Experimental): All participants randomly assigned to the intervention group will receive free near or distance vision correction glasses based on their refractive error. Participants can choose from a variety of frames, and the research team will customize the glasses according to their pupillary distance and prescription. Once the glasses are ready, they will be provided to the participants following standard usage instructions. In case of loss or damage, participants should report it to the project team and will be provided with replacement glasses as needed. Each year, participants in the intervention group will undergo an eye exam to assess changes in vision, and their glasses prescription will be updated if necessary.
  Interventions: Device: Free Prescription Glasses
- Prescription-Only Control group (No Intervention): All participants randomly assigned to the control group will receive an eyeglass prescription, but free glasses will not be provided during the study. At the end of the study, the research team will provide near or distance vision correction glasses free of charge based on the needs of the control group participants.

INTERVENTIONS:
Device: Free Prescription Glasses — Participants can choose from a variety of frames, and the research team will customize the glasses according to their pupillary distance and prescription. Once the glasses are ready, they will be provided to the participants following standard usage instructions. In case of loss or damage, participants should report it to the project team and will be provided with replacement glasses as needed. Each year, participants in the intervention group will undergo an eye exam to assess changes in vision, and their glasses prescription will be updated if necessary.
  Arms: Free Prescription Glasses Intervention group

SUMMARY:
The aim of this project is to explore whether vision correction can effectively slow cognitive decline in older adults.

The primary question it seeks to answer is: Can providing free near and/or distance vision correction glasses to older adults with refractive errors or uncorrected vision, who have normal baseline cognition and hearing, reduce the rate of cognitive decline over 36 months in a cost-effective manner? Researchers will compare the rate of cognitive decline over 36 months between older adults who receive refractive correction and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Older adults who meet all of the following criteria will be eligible to participate in this study:

  * Registered as a rural resident (holding rural household registration);
  * Age from 60 to 79 years at the time of enumeration;
  * Resident in the household for > = 3 months and planning to reside in the local area for the trial duration;
  * Distance vision impairment (VI, presenting visual acuity [VA] < 6/18 in the better-seeing eye and improving to > = 6/18 with spectacles) and/or near VI (presenting near vision < N6 at 40 cm and improving to > = N6 with spectacles);
  * Independent mobility with or without the support of a walking stick;
  * Chinese version of the Mini-Mental State Examination (C-MMSE) score above the following cut-offs (out of 30): >17 for illiterate participants, >20 for those with primary school education, >22 for those with junior high school education, and >23 for those with high school education or above.
  * Willingness to participate, to be randomized to either study group, and to adhere to the protocol

Exclusion Criteria:

* Presence of glaucoma or visually significant cataract, or a history of surgical treatment for these or other major ocular conditions;
* Consistent use of prescription spectacles and/or hearing aids;
* Serious medical illness likely to result in loss to follow-up. Those less severely affected by conditions such as hypertension and/or diabetes will be eligible;
* Failure on the whispered voice hearing screening test in the better ear (unable to repeat > = 3 out of 6 words whispered from behind the participant at a distance of 50 cm);

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 964 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
**Chinese version of the Global Cognitive Score Scale** | Each participant will undergo cognitive assessments at baseline, 12 months, 24 months, and 36 months to evaluate the impact of the intervention on cognitive decline.
  The primary endpoint is the change in cognitive function over three years, which is comprehensively determined using the Chinese version of the Global Cognitive Score Scale-by administering the Chinese version Mini-Mental State Examination (C-MMSE), Beijing version of the Montreal Cognitive Assessment (MoCA), Telephone Interview for Cognitive Status (TICS), Community Screening Instrument for Dementia Interviewee Part (CSI-D), and Number Series Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Community health service centers, Ya'an, Sichuan, China